CLINICAL TRIAL: NCT05578716
Title: GRANDIOSA - Growth, Allergy and Neurodevelopment in Infants on Hydrolysed Formula
Brief Title: Growth, Allergy and Neurodevelopment in Infants on Hydrolysed Formula
Acronym: GRANDIOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Lund University (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Magnus Domellöf, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20210707401
Record Dates: First submitted 2022-09-19; First posted 2022-10-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Infant Formula
Keywords: Infant nutrition; Food hypersensitivity; Dermatitis, Atopic; Protein hydrolysates; Spectroscopy, Near-Infrared
MeSH Terms: conditions — Food Hypersensitivity; Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either standard formula or one of two partially hydrolysed study formulae. Included in the study will also be a group of breast-fed infants acting as reference group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each formula in the study will have the same packaging besides from colour coding (green, blue, yellow). None of the study personnel are aware of which colour represents which formulae during the course of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study formula 1 (Experimental): Formula-fed intervention group randomised to one of two study formulae
  Interventions: Dietary Supplement: Partially hydrolysed formula
- Study formula 2 (Experimental): Formula-fed intervention group randomised to one of two study formulae
  Interventions: Dietary Supplement: Partially hydrolysed formula
- Standard formula (No Intervention): Formula-fed control group randomised to standard formula
- Breast feeding (No Intervention): Reference group with exclusively breast-fed infants

INTERVENTIONS:
Dietary Supplement: Partially hydrolysed formula — Partially hydrolysed formula
  Arms: Study formula 1; Study formula 2

SUMMARY:
Breastfeeding is the recommended diet for all infants during the first half of infancy and is associated with numerous health benefits. However, when breastfeeding is not possible, an infant formula is the only nutritive alternative. Formula-fed infants have a different growth pattern compared to breastfed infants. Studies have shown that the higher protein content in infant formula compared to breastmilk results in a more rapid weight gain and an increased risk of overweight and obesity in childhood. For this reason, both quantity and quality of protein in infant formulae have been optimized during the last decade, to better meet the needs of infants and to support growth close to that of breastfed infants.

Protein hydrolysis, a common modification of infant formulae, has originally been developed for treatment of cow's milk protein allergy. Certain hydrolysed formulae have been suggested to prevent atopic eczema when given to infants with a family history of allergic disease but as of yet, the allergy preventive effect in infants without increased risk of allergic disease has been little studied. Partially hydrolysed infant formulae have also been suggested to reduce common functional gastrointestinal symptoms in infants.

New protein hydrolysates are continually developed for use in infant formulae, with the aim of reducing allergenicity, while ensuring optimal growth and development of infants. It is important to study the effects on growth and health outcomes in infants who are fed formulae based on these newly developed hydrolysates as compared to those fed standard intact protein formulae or breastmilk.

The overall aims of the current study are to evaluate the effects of two new hydrolysates on growth, immunological biomarkers, neurodevelopment, protein metabolism and gut microbiota in a randomized, controlled clinical trial of healthy infants. In compliance with European Food Safety Authority (EFSA) regulations for novel infant formulas based on hydrolysed protein, the primary outcome is change in weight standard deviation score (SDS) from baseline until 5 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants born at term
* Birth weight 2500 to 4500 gram
* Either exclusive breast-feeding (reference group) or exclusive formula-feeding (intervention and control group)

Exclusion Criteria:

* Suspected or verified food allergy
* Suspected or verified infant colic

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Weight | At 5 months of age
  Primary outcome is weight Standard Deviation Score (SDS) at the end of the intervention.

SECONDARY OUTCOMES:
Length. | At enrollment at 2 months of age and monthly during the intervention up to 5 months of age.
  Growth pattern during the course of the intervention measured by length in centimeters and SDS.
Head circumference. | At enrollment at 2 months of age and monthly during the intervention up to 5 months of age.
  Growth pattern during the course of the intervention measured by head circumference in centimeters and SDS.
Body composition | At 4 months of age
  Assessing differences in body composition between study groups using fat percentage as measured by PeaPod (Pletysmography).
Gastrointestinal tolerance. | At enrollment at 2 months of age and during the intervention up to 5 months of age.
  Gastrointestinal tolerance using diary for information about stool frequency and consistency (in four grades from diarrhea to hard stools) in combination with questionnaire filled in by the parents based on Rome IV criteria for functional gastrointestinal disorders.
Gastrointestinal immunology. | At enrollment at 2 months of age and during the intervention up to 5 months of age.
  Markers of gastrointestinal immune activation using analysis of calprotectin, eosinophilic derived neurotoxin and secretory Immunoglobulin A (IgA) in fecal samples.
Eczema severity, parent report. | At enrollment at 2 months of age and during the intervention up to 5 months of age.
  Parents will fill in the Patient-Oriented Eczema Measure (POEM) score monthly during the intervention.
Eczema severity, clinical assessment. | At enrollment at 2 months of age and during the intervention up to 5 months of age.
  Excema severity is assessed at every study visit using the Eczema Area and Severity Index (EASI).
Allergy. | At enrollment at 2 months of age and at the end of the intervention at 5 months of age.
  Sensitization to cow's milk protein is assessed by Immunoglobulin E (IgE) in serum using ImmunoCap.
Immunologic activity. | At enrollment at 2 months of age and at the end of the intervention at 5 months of age.
  Blood cytokine patterns using Luminex: Interleukin 2 (IL-2) as a marker of general T cell activity. Interferon gamma (IFN-γ) as a marker of Helper T cells type 1 (Th1) activity. Interleukin 4 (IL-4) as a marker of helper T cells type 2 (Th2) activity. Tumor growth factor beta type 1 (TGF-β1) as a marker of T cell regulatory activity. Interleukin 17 A (IL17-A) as a marker of helper T cell type 17 (Th17) activity. C reactive protein (CRP) in plasma as a marker of general inflammatory response.
Metabolic biomarkers in blood. | At enrollment at 2 months of age and at the end of the intervention at 5 months of age.
  Insulin-like growth factor-1 (IGF-1). Insulin. C-peptide. Leptin. Leptin-receptor.
Markers of protein metabolism. | At enrollment at 2 months of age and at the end of the intervention at 5 months of age.
  Plasma amino acids. Blood urea nitrogen.
Microbiota | At enrollment at 2 months of age and during the intervention up to 5 months of age.
  Composition and diversity of the gut microbiota analysed in fecal samples. Bacterial DNA will be extracted and the V3-V4 region of the 16S rRNA gene will be amplified. Sequencing of all samples takes place on the Illumina MiSeq platform. Based on the results, we will also use metagenomic or Nanopore sequencing for deeper characterization of microbial composition and functions.
Neurodevelopment at 6 months of age. | At 6 months of age.
  Response in cerebral blood flow to visual and auditory stimuli as measured by functional near-infrared spectroscopy (fNIRS).
Neurodevelopment at 12 months of age. | At 12 months of age.
  Bayely scales of infant development (BSID) 3rd edition. Higher score is interpreted as better outcome.
Neurodevelopment at 3 years of age. | At 3 years of age
  Wechsler Preschool and Primary Scale of Intelligence (WIPPSI) 4th edition. Higher score is interpreted as better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Domellöf, MD, PhD, Principal Investigator — Department of Clinical Sciences, Pediatrics, Umeå University Hospital
Locations (2):
- Sweden (2):
  - Department of clinical science, Preventive Paediatrics, Lund university, Malmo
  - Department of Clinical Sciences, Pediatrics, Umeå University Hospital, Umeå